CLINICAL TRIAL: NCT05416060
Title: Dulce Digital 2.0 - Innovative Diabetes Self-Management in the Digital Age
Acronym: Dulce Digital
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Whittier Diabetes Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MISP-60691; MISP-60691 (Other Grant/Funding Number: Merck)
Record Dates: First submitted 2022-06-06; First posted 2022-06-13 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Type 2
Keywords: Diabetes; Health Education; mHealth Technology; Group Education; Telehealth; Text-Based
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Health Education

STUDY DESIGN:
Intervention Model Description: This is a three-arm, non-blinded, randomized, controlled, parallel-groups, comparative effectiveness trial with N=150 participants.
  The protocol was developed in accordance with Good Clinical Practice, SPIRIT, and CONSORT 2013 guidelines.
Who Masked: Outcomes Assessor
Masking Description: This is a three-arm, non-blinded, randomized, controlled, parallel-groups, comparative effectiveness trial with N=150 participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dulce Digital (Experimental): Patients will participate in a text-based diabetes self-management educational and support (DSME/S) program and receive ongoing support via text messages designed to improve knowledge, health beliefs, self-management behaviors and clinical outcomes.
  Interventions: Behavioral: Dulce Digital Text-Based Education
- Project Dulce Telehealth DSME/S (Experimental): Patients will participate in live a peer-led Telehealth diabetes self-management education and support program.
  Interventions: Behavioral: Project Dulce Telehealth
- Project Dulce Live DSME/S (Experimental): Patients will participate in live a peer-led Telehealth diabetes self-management education and support program.
  Interventions: Behavioral: Project Dulce Live

INTERVENTIONS:
Behavioral: Dulce Digital Text-Based Education — Participants will be enrolled in the digital texting platform, Dulce Digital in which they will receive on-going support via text messages for 6 months, derived from the Project Dulce curriculum. Topics include medication reminders, motivational prompts, nutrition and stress reduction tips and request to submit weekly blood glucose numbers.
  Arms: Dulce Digital
Behavioral: Project Dulce Telehealth — Project Dulce will consist of a group-based telehealth diabetes self-management education program consisting of a 5 -week curriculum delivered by a peer educator in English or Spanish. The curriculum provides skills and tools needed to adapt to a life with diabetes and change behaviors. The curriculum covers diabetes and its complications, the role of diet, exercise, and medication, and the importance of self-monitoring. It is presented over 5 weeks where participants learn and practice self-management skills, and help one another address family, cultural or health system barriers to managing your diabetes.
  Arms: Project Dulce Telehealth DSME/S
Behavioral: Project Dulce Live — Project Dulce will consist of a group-based diabetes self-management education program consisting of a 5 -week curriculum delivered by a peer educator in English or Spanish. The curriculum provides skills and tools needed to adapt to a life with diabetes and change behaviors. The curriculum covers diabetes and its complications, the role of diet, exercise, and medication, and the importance of self-monitoring. It is presented over 5 weeks where participants learn and practice self-management skills, and help one another address family, cultural or health system barriers to managing your diabetes.
  Arms: Project Dulce Live DSME/S

SUMMARY:
The proposed research, "Dulce Digital 2.0," will evaluate two mHealth adaptions of Project Dulce that are designed to improve digital health literacy, increase underserved individuals' capacity to access and engage with vital digital health information, and in turn, improve clinical and behavioral outcomes in at-risk adults with diabetes. Expanding access to care in populations faced with challenges of low socioeconomic status and health literacy is a step toward reducing health disparities and positively affecting care. The literature shows that identifying which groups of participants are most likely to benefit from telehealth interventions is an important factor in improving the evidence base for digital health literacy. Dulce Digital 2.0 is highly scalable once the technical infrastructure is built. More importantly, by helping to reduce existing inequities in access to diabetes care and accurate digital health information the model could help to improve health outcomes on a larger scale. The use of digital technology in the delivery of healthcare interventions is increasingly common. Barriers to engagement in digital technology exist among those in underserved populations due to language, access to equipment and internet, education level, exposure to and comfort with technology, and pre-existing deficits in health literacy. The proposed research will investigate the effectiveness of two digital approaches to improving the self-management and digital health skills of underserved participants with diabetes compared to tradition in-person self-management education: 1) live self-management education, traditional in-person classes; 2) live self-management education using a telehealth distance learning platform; and 3) a series of text-based messages, not requiring a smart phone or internet connection, that encourage healthy self-management behaviors.

DETAILED DESCRIPTION:
Diabetes self-management education using digital platforms including, telehealth group visits, text-based messages and live delivery will result in improvements in diabetes health behaviors, patient engagement, health literacy and HbA1c.

Diabetes disproportionately affects racial and ethnic communities. The investigator developed Project Dulce, an American Diabetes Association-recognized and Medicare-approved Diabetes Self-Management Education and Support (DSME/S) program addresses the needs of a racially and ethnically diverse San Diego population and includes a multi-disciplinary team with peer educators delivering DSME/S. Previous trials have shown Project Dulce team-care improves clinical management and reduces costs and that the peer education alone improves clinical outcomes in Hispanics with Type 2 Diabetes across 10 months.

Mobile health (mHealth) technologies represent a viable way to overcome many of these barriers and extend the reach of DSME/S to participants who need it most.

During the coronavirus disease (COVID-19) pandemic, Project Dulce was adapted for group telehealth settings and delivered via the electronic medical record (EMR) scheduling system. Additionally, a previously developed text messaging platform-Dulce Digital was offered to extend the reach of the care team through educational and motivational messaging, medication reminders, and blood glucose monitoring prompts. A previous randomized controlled trial of Dulce Digital demonstrated a significant reduction of HbA1c across 10 months versus usual care in Hispanics with diabetes. While live Project Dulce and Dulce Digital programs have demonstrated improvements in clinical and cost outcomes in Hispanic patients, a comparative analysis of live, group telehealth and text messaging programs has not been done. This study will assess a direct comparison of each of these modalities to explore the feasibility, acceptance, and effectiveness of each delivery modality across Hispanic communities living with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic/Latino adults who are registered patients of Scripps Health
* Diagnosis of Type 2 Diabetes
* HbA1c greater than or equal to 8% within the last 60 days

Exclusion Criteria:

* Severe illness precluding visits to clinic
* Liver function tests (ALT and AST) > 3 times the upper limit of normal
* Body mass index ≤ 23 kg/cm
* History of malignancy, except subjects who have been disease-free for >2 years, or whose only malignancy has been basal or squamous cell skin carcinoma
* Creatinine >3.5
* History of drug or alcohol abuse within 12 months prior to randomization
* Current enrollee in DSME/S
* Blood donation of one pint or more within the past 30 days, or plasma donation within 7 days prior to screening
* Anemia
* Lack of minimal literacy needed to participate in the text intervention
* Severe auditory or visual problems
* Primary language other than Spanish or English
* Not willing to carry a mobile phone
* Pregnant
* Plans to relocate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Baseline Glycosylated Hemoglobin A1C (HbA1c) at 3 months | 3 months
  Change in Baseline Glycosylated Hemoglobin A1C (HbA1c) at 3 months; % Units HbA1c is measure of blood sugar level and assessed using blood samples following a 12-hour fast. Samples will be process by Quest Diagnostics Inc and assayed by Immunoturbidimetry (integra 800, Roche). Higher is worse.
Change from Baseline in Baseline Glycosylated Hemoglobin A1C (HbA1c) at 6 months | 6 months
  Change in Baseline Glycosylated Hemoglobin A1C (HbA1c) at 6 months; % Units HbA1c is measure of blood sugar level and assessed using blood samples following a 12-hour fast. Samples will be process by Quest Diagnostics Inc and assayed by Immunoturbidimetry (integra 800, Roche). Higher is worse.

SECONDARY OUTCOMES:
Change from Baseline Diabetes Distress (DDS-17) at 3 months | 3 months
  The Diabetes Distress Scale (DDS-17) is a self-report instrument for adults with type 2 diabetes. The scaled yields an overall distress score based on the average of response on the 1-6 scale for all 17 items. The DDS-17 identifies three levels of specificity of diabetes distress information for use in clinical care, from overall emotional distress related to diabetes to highly specific sources of diabetes distress. Higher score is worse.
Change from Baseline Diabetes Distress (DDS-17) at 6 months | 6 months
  The Diabetes Distress Scale (DDS-17) is a self-report instrument for adults with type 2 diabetes. The scaled yields an overall distress score based on the average of response on the 1-6 scale for all 17 items. The DDS-17 identifies three levels of specificity of diabetes distress information for use in clinical care, from overall emotional distress related to diabetes to highly specific sources of diabetes distress.
Change from Baseline Diabetes Treatment Satisfaction Questionnaire (DTSQ) at 3 months | 3 months
  The DTSQ scale has been shown to be useful in clinical trials evaluation of new technologies and has been used as one outcome indicator in routine audit diabetes care. It is composed of 8 questions, scored by patients on a scale ranging from 0 ("very dissatisfied", "very inconvenient") to 6 ("very satisfied", "very convenient"). It is composed of 2 factors. The first factor assesses treatment satisfaction (6 questions). These questions ask about "satisfaction with current treatment", "flexibility", "convenience", "understanding of diabetes", "recommend treatment to others" and "willingness to continue", respectively. The second factor (2 questions) which assess the burden from hyper- and hypoglycemia, respectively (0 "none of the time" to 6 "most of the time"). Treatment satisfaction is assessed as the sum of scores of 6 questions on the first factor (total score 36). A higher score indicates higher treatment satisfaction.
Change from Baseline Diabetes Treatment Satisfaction Questionnaire (DTSQ) at 6 months | 6 months
  The DTSQ scale has been shown to be useful in clinical trials evaluation of new technologies and has been used as one outcome indicator in routine audit diabetes care. It is composed of 8 questions, scored by patients on a scale ranging from 0 ("very dissatisfied", "very inconvenient") to 6 ("very satisfied", "very convenient"). It is composed of 2 factors. The first factor assesses treatment satisfaction (6 questions). These questions ask about "satisfaction with current treatment", "flexibility", "convenience", "understanding of diabetes", "recommend treatment to others" and "willingness to continue", respectively. The second factor (2 questions) which assess the burden from hyper- and hypoglycemia, respectively (0 "none of the time" to 6 "most of the time"). Treatment satisfaction is assessed as the sum of scores of 6 questions on the first factor (total score 36). A higher score indicates higher treatment satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Athena Philis-Tsimikas, MD, Principal Investigator — Scripps Health
Locations (2):
- United States (2):
  - Scripps Chula Vista Diabetes Center, Chula Vista, California
  - Scripps Whittier Diabetes Institute, San Diego, California

IPD SHARING:
Plan to Share IPD: No